CLINICAL TRIAL: NCT03252639
Title: A Prospective Study of Using Parenchymal Blood Volume(PBV) for Endovascular Treatment of Renal Arterial Stenosis
Brief Title: A Study of Using Parenchymal Blood Volume(PBV) for Endovascular Treatment of Renal Arterial Stenosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-2016-1.20
Record Dates: First submitted 2017-08-10; First posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Renal Artery Stenosis; Renal Blood Perfusion
Keywords: Renal Artery Stenosis; Renal Blood Perfusion
MeSH Terms: conditions — Renal Artery Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Renal Artery Stenosis: Patients with renal artery stenosis which may benefit from endovascular treatment will be recruited. Those patients who cannot benefit from this procedure will be excluded.
  Interventions: Procedure: EVT for RAS & PBV acquisition protocol for target kidneys

INTERVENTIONS:
Procedure: EVT for RAS & PBV acquisition protocol for target kidneys

SUMMARY:
This study will use PBV technique to quantitatively assess the improvement of renal perfusion before and after endovascular treatment (EVT) of renal artery stenosis.

DETAILED DESCRIPTION:
BACKGROUND: Renal artery stenosis (RAS) is one of the main reasons for secondary hypertension and renal failure, which etiologies include atherosclerosis, fibromuscular dysplasia and takayasu arteritis. Endovascular treatment under digital subtraction angiography (DSA) is an option to treat this disease. However, the technical success of this procedure is mainly based on morphology of its targeting renal artery without any quantified data towards renal blood perfusion. Thus, this study will try to solve how renal blood perfusion changes before and after endovascular treatment of renal artery stenosis.

DESIGN NARRATIVE:

This prospective cohort study will recruit patients with renal artery stenosis. PBV data will be obtained before and after their endovascular treatments. The volume of target kidney and its mean density of contrast from PBV data will be calculated as indicators for renal perfusion. And the relation between the percentage of stenosis and renal perfusion will be analyzed. The follow-up will last for one year. At 6-month and 12-month follow-up, DSA and PBV acquisition protocol will be undertaken again to evaluate renal blood perfusion in the long term.

ELIGIBILITY:
Inclusion Criteria:

Patients should meet all of the following criteria:

1. Age ≥ 18.
2. Renal artery stenosis is greater than or equal to 80% and less than 100% by duplex, CT angiography or magnetic resonance angiography.
3. The target kidney remains functional(tested by radionuclide imaging)
4. Documented history of hypertension on two or more anti-hypertensive medications OR estimated glomerular filtration rate (eGFR) less than 60 mL per minute per 1.73 m^2, calculated by the modified Modification of Diet in Renal Disease formula.
5. The length of target kidney is >8cm.

Exclusion Criteria:

Patients meet any of the following criteria should be excluded.

1. Unable or willing to comply with study protocol or procedures.
2. Pregnancy or lactation.
3. History of kidney transplant.
4. Currently in acute pulmonary edema OR systolic ejection fraction of heart <30% OR respiratory failure due to hypertension or acute coronary syndrome or cerebrovascular accident in past 3 months.
5. The eGFR is less than 15 mL per minute per 1.73 m^2 OR serum Cr is greater than 3.0 mg/dl on the day of randomization.
6. Other known reason nonischemic kidney injure(e.g. nephritis). If it is diabetic nephropathy, 24h urinary protein should be more then 3g.
7. Aorta has stenosis(greater than 30%).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who meet the inclusion criteria, are willing to join this trial and treated in the department of vascular surgery, Peking Union Medical College Hospital will be included in this prospective cohort study.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Kidney Volume | 15 minutes before endovascular treatment, changes at 15 minutes after endovascular treatment, 6-month and 12-month follow-up respectively.
  the volume of kidney, which is able to indicate total blood volume of kidney, in target kidney
mean density of contrast | 15 minutes before endovascular treatment, changes at 15 minutes after endovascular treatment, 6-month and 12-month follow-up respectively.
  the mean density of contrast, which is able to represent renal blood perfusion, in target kidney

CONTACTS AND LOCATIONS:
Overall Officials: Bao Liu, MD, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No